CLINICAL TRIAL: NCT00156975
Title: Adjuvant Chemotherapy With Oxaliplatin and Capecitabine Versus Follow-up After Resection of Colorectal Liver Metastases- Randomized Phase III Study
Brief Title: Oxaliplatin and Capecitabine Versus Follow-up After Resection of Colorectal Liver Metastases
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arbeitsgruppe Lebermetastasen und Tumoren (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADHOC
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2007-04

CONDITIONS: Colorectal Neoplasms; Liver Metastases
Keywords: Oxaliplatin; Capecitabine; Chemotherapy; Resection; Liver metastases; Liver resection; Adjuvant
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine
Drug: Oxaliplatin

SUMMARY:
Primary endpoint of the study is to prove the superiority of an adjuvant therapy with oxaliplatin/ capecitabine until the first occurrence of appearance of a tumour. Occurrences in the meaning of this study are the appearance of a relapse of the tumour, of metastases, of a second tumour or death of any reason.

DETAILED DESCRIPTION:
Prospective, randomized, multi-centre, open phase III study with two parallel groups of patients according to the eligibility criteria. The times in both hierarchical classified endpoints will be measured as times from randomization.

Patients with macroscopic complete resection of colorectal liver metastases will be randomized in:

Arm A: post-operative adjuvant therapy with Capecitabine/ Oxaliplatin over 6 months and follow-up

or

Arm B: follow-up

Randomization: stratification after Scores of Fong et al:

* number of metastases (1 vs. >=1)
* maximal diameter of the metastasis (<= 5cm vs. > 5cm)
* disease free interval (>= 12 months vs. > 12 months)
* CEA (<= 200ng/l vs. >200 ng/l) in the strata 0-1, 2 and >= 3,

ELIGIBILITY:
Inclusion Criteria:

* patients after R0-resection of colorectal liver metastases
* age: >= 18 years
* Karnofsky-Index >= 70%
* neutrophiles >1,5 x10e9/l, thrombocytes 100 x10e9/l
* adequate contraception for male and female patients
* oral and written informed consent (GCP)

Exclusion Criteria:

* other prior malignancies, except treated in situ-carcinoma of cervix or tumours of skin without indication to a melanoma (or 10 years tumourfree)
* other participation in clinical trials within 30 days before randomization
* previous chemotherapy (except adjuvant chemotherapy with an interval of >= 6 months)
* creatinine clearance <50 ml/min
* hepatic insufficiency (ALAT, ASAT, Bilirubin, AP >5 x upper limit)
* peripheral neuropathy > CTC grade 1
* uncontrolled cardiac insufficiency or angina pectoris
* active infections
* severe neurological or psychiatric illness
* breast-feeding or pregnant women
* incapacity to take part in regular visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384
Dates: Start 2004-11

PRIMARY OUTCOMES:
Primary outcomes:
Disease free survival

SECONDARY OUTCOMES:
Secondary outcomes:overall survival,acute- and longtime toxicity of chemotherapy, molecular predictive markers for the risk of relapse and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Wolf O. Bechstein, Prof. Dr., Principal Investigator — Arbeitsgruppe Lebermetastasen und Tumoren
Locations (3):
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus, Medizinische Klinik, Dresden, Saxony
  - Universitaetsklinikum Essen, Klinik für Allgemein- und Transplantationschirurgie OPZ II, Essen
  - Klinik für Allgemein- und Gefäßchirurgie , J. W. Goethe Universität, Frankfurt am Main